CLINICAL TRIAL: NCT02717312
Title: Defect in Cesarean Scar: A Prospective Study of Prevalence, Risk Factors and Impact on Menstrual Disorders and Quality of Life
Brief Title: Prevalence, Risk Factors and Consequences Related to Cesarean Scar Defect (Defect in Cesarean Scar)
Acronym: DICE
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: City of Tampere (Unknown); Finnish Medical Foundation (Network); Competitive State Research Funding of Tampere University Hospital (Unknown); Tampere University Hospital Support Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: R15104
Record Dates: First submitted 2016-03-09; First posted 2016-03-23 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Cesarean Scar Defect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The rates of cesarean section (CS) are rising all over the world. Worldwide the number of CS is millions every year. CS is one of the most frequently performed operation for women. As a consequence many women have a scar in their uterus. Cesarean scar may be associated with complications in later pregnancies. In recent years there have also been a few reports indicating that cesarean scar could potentially be associated with menstrual disorders and infertility. The impact of cesarean scar defect on long term welfare or quality of life is not clear.

In some women with a history of CS it is possible to recognise a defect in the site of previous uterotomy years after the performed CS by sonographic examination. This defect in the scar, also called as a niche, is a consequence of incomplete healing of the scar in the lower part of uterus. To date there is uncertainty relating to the factors that lead to poor healing of cesarean scar. Also impact of cesarean scar defect on later well-being and later pregnancies are not properly known.

The purpose of this study is to investigate the prevalence and the risk factors of cesarean scar defect. Also the impact of cesarean scar defect on women´s menstrual health, fertility, further deliveries and quality of life will be investigated.

This study is a prospective observational cohort study. Women at the age of 18-45 years who will give birth by elective or emergency CS will be asked to participate. Women are recruited within two days of CS. Women with known uterus anomaly or von Willebrand disease will be excluded.

The prevalence of scar defect will be evaluated by transvaginal sonography and contrast-enhanced sonohysterography using saline infusion. Both 2-dimensional and 3-dimensional sonography will be used. Sonographic evaluation will take place 6 months after the CS.

The following definition for CS scar defect will be used: myometrial discontinuity with a depth of ≥2 mm at the site of cesarean scar that communicates with the uterine or cervical cavity as seen on transvaginal sonography with or without saline infusion.

The prevalence of menstrual disorders will be evaluated 12 months after the CS. The subjects will be asked to report the number of menstrual bleeding days once a month during 3 consecutive months. Postmenstrual spotting is defined as ≥2 days of brownish discharge at the end of menstruation with total bleeding days of ≥7 or non-cyclic bleeding not related to menstruation.

ELIGIBILITY:
Inclusion Criteria:

* Women who gives birth by cesarean section whether it will be an elective surgery or an emergency surgery during labour

Exclusion Criteria:

* Uterus anomaly or von Willebrand disease
* Informed consent not provided

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women undergoing cesarean section
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Association between cesarean scar defect and post menstrual spotting | 15 months
  Postmenstrual spotting is defined as ≥2 days of brownish discharge at the end of menstrual bleeding with total bleeding days ≥7 or inter menstrual non-cyclic bleeding not related to menstruation.

SECONDARY OUTCOMES:
Quality of life related to cesarean scar defect | 10 years
  Quality of life related to cesarean scar defect will be assessed by using rand36 score.
Association between cesarean scar and adverse pregnancy outcome | 10 years
  Adverse pregnancy outcome includes spontaneous abortion, cesarean scar pregnancy, uterine rupture in later pregnancy and the rate of vaginal birth/cesarean section in later pregnancies.
Prevalence of cesarean scar defect measured by sonography | 6 months
  Number of participants with cesarean scar defect. Cesarean scar defect is defined as myometrial discontinuity with a depth of ≥2 mm at the site of cesarean scar that communicates with the uterine or cervical cavity as seen on transvaginal sonography with or without saline infusion.
Impact of cervical opening at the time of cesarean section on the prevalence of cesarean scar defect. | 6 months
  Association between cervical opening at the time of operation (cm) and detected cesarean scar defect (6 months after the operation).

CONTACTS AND LOCATIONS:
Overall Officials: Synnöve Staff, MC PhD, Study Director — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No